CLINICAL TRIAL: NCT04856319
Title: The Effect of Pre-operative Single Dose Antibiotic Prophylaxis on the Post-operative Implant Success
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Mustafa YILMAZ, Assist Prof, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Implant prophylaxis
Record Dates: First submitted 2021-04-12; First posted 2021-04-23 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Tooth Loss
Keywords: Dental Implants; Antibiotic Prophylaxis
MeSH Terms: conditions — Tooth Loss | interventions — Antibiotic Prophylaxis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The patients and the surgeon will be masked if antibiotics or placebo were used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylaxis (Active Comparator): 2 g amoxicillin+clavulanic acid 1 hour prior to dental implant surgery
  Interventions: Procedure: Dental implant placement; Drug: Antibiotic prophylaxis
- Placebo (Placebo Comparator): placebo 1 hour prior to dental implant surgery
  Interventions: Procedure: Dental implant placement; Other: Placebo

INTERVENTIONS:
Procedure: Dental implant placement — Insertion of not more than two dental implants at the same area
Drug: Antibiotic prophylaxis — Per-os 2g amoxicillin+clavulanic acid will be administered one hour prior to the surgery
  Arms: Prophylaxis
Other: Placebo — Per-os placebo (inert polysaccharide) will be administered one hour prior to the surgery
  Arms: Placebo

SUMMARY:
There is no consensus on antibiotic prophylaxis in dental implant applications, and its necessity is controversial. Current reports on antibiotic use are insufficient. Also, other than antibiotic prophylaxis, data that may affect the post-operative situation such as the patient's gender, age, smoking, duration of surgery, length of the operation field, flap design have not been evaluated comprehensively.

This study aims to evaluate post-operative complications, implant success, and implant stability in 50 individuals: preoperative single dose of 2 g amoxicillin + clavulanic acid (25) and placebo (25).

ELIGIBILITY:
Inclusion Criteria:

* Tooth loss

Exclusion Criteria:

* Systemic disease
* Lactation/pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Baseline implant stability / osseointegration | Baseline
  Periotest M
10th day implant stability / osseointegration | 10th day
  Periotest M
1st month implant stability / osseointegration | 1st month
  Periotest M
Final implant stability / osseointegration | 3rd month
  Periotest M
Radiographic bone loss | 3rd month
  The distance of the bone crest to the implant shoulder
Early healing index (Wachtel et al) | 10th day
  Complete flap closure (1), fine fibrin line (2), fibrin clot (3), partial necrosis (4), complete necrosis (5)
Early healing index (Wachtel et al) | 1st month
  Complete flap closure (1), fine fibrin line (2), fibrin clot (3), partial necrosis (4), complete necrosis (5)

SECONDARY OUTCOMES:
Operation duration | Baseline
  Duration between the first incision and the last suture
Painkiller (0-3 days) | Baseline - 3rd day
  500 mg paracetamol, the count of the painkillers the subject used
Painkiller (3-10 days) | 3rd day - 10th day
  500 mg paracetamol, the count of the painkillers the subject used
Operation zone length | Baseline
  (mm) the crestal incision and vertical incision (if applied) length

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Yılmaz, PhD, Principal Investigator — Biruni University, assistant professor
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be shared
Supporting Information: Study Protocol
Time Frame: Starting one year after the publication
Access Criteria: All the collected data will be accessible to researchers conducting meta-analysis or examining the reliability of our study